CLINICAL TRIAL: NCT01089270
Title: Ioflupane I123 (DaTSCAN) and Positron Emission Tomography-computed Tomography Fludeoxyglucose (PET-CT FDG) to Assess Brain Function of Parkinson Patients' First Degree Relatives
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Einat Even-Sapir MD, PhD. Head, Dept of Nuclear Medicine, Tel Aviv Sourasky Medical Center
Other Study IDs: TASMC-10-EES-0519-CTIL
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson; fdg pet-ct; i123 dat scan; first degree relatives of diagnosed Parkinson patients; with no clinical evidence of movement disorders
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Parkinson Disease is one of the most common neurodegenerative illnesses. First degree relatives of Parkinson patient are in high risk for developing the disease. We will try to detect early changes in brain metabolism before the appearance of Parkinson symptoms.

Participants: first degree relatives of diagnosed Parkinson patients that carry a gene mutation in either LRRK2 or GBA genes.

The examination results will be given to the participants by a doctor from the neurology department.

ELIGIBILITY:
Inclusion Criteria:

* healthy first degree relatives of diagnosed Parkinson patients

Exclusion Criteria:

* patients unable to understand and sign an informed consent
* minors
* people with psychiatric disorders or a history of major head trauma

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First degree relatives of diagnosed Parkinson patients that carry either LRRK2 or GBA gene mutation.
  Ages: 30-80
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Einat Even-Sapir, MD, PhD, Principal Investigator — Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
Locations (1):
- Department of Nuclear Medicine, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Volkow ND, Ding YS, Fowler JS, Wang GJ, Logan J, Gatley SJ, Hitzemann R, Smith G, Fields SD, Gur R. Dopamine transporters decrease with age. J Nucl Med. 1996 Apr;37(4):554-9. PMID 8691238
- [Background] Huang Y, Cheung L, Rowe D, Halliday G. Genetic contributions to Parkinson's disease. Brain Res Brain Res Rev. 2004 Aug;46(1):44-70. doi: 10.1016/j.brainresrev.2004.04.007. PMID 15297154
- [Background] Vila M, Przedborski S. Genetic clues to the pathogenesis of Parkinson's disease. Nat Med. 2004 Jul;10 Suppl:S58-62. doi: 10.1038/nm1068. PMID 15272270
- [Background] von Bohlen und Halbach O, Schober A, Krieglstein K. Genes, proteins, and neurotoxins involved in Parkinson's disease. Prog Neurobiol. 2004 Jun;73(3):151-77. doi: 10.1016/j.pneurobio.2004.05.002. PMID 15236834
- [Background] Farrer M, Stone J, Mata IF, Lincoln S, Kachergus J, Hulihan M, Strain KJ, Maraganore DM. LRRK2 mutations in Parkinson disease. Neurology. 2005 Sep 13;65(5):738-40. doi: 10.1212/01.wnl.0000169023.51764.b0. PMID 16157908
- [Background] Orr-Urtreger A, Shifrin C, Rozovski U, Rosner S, Bercovich D, Gurevich T, Yagev-More H, Bar-Shira A, Giladi N. The LRRK2 G2019S mutation in Ashkenazi Jews with Parkinson disease: is there a gender effect? Neurology. 2007 Oct 16;69(16):1595-602. doi: 10.1212/01.wnl.0000277637.33328.d8. PMID 17938369
- [Background] Herholz K, Heiss WD. Positron emission tomography in clinical neurology. Mol Imaging Biol. 2004 Jul-Aug;6(4):239-69. doi: 10.1016/j.mibio.2004.05.002. PMID 15262239
- [Derived] Artzi M, Even-Sapir E, Lerman Shacham H, Thaler A, Urterger AO, Bressman S, Marder K, Hendler T, Giladi N, Ben Bashat D, Mirelman A. DaT-SPECT assessment depicts dopamine depletion among asymptomatic G2019S LRRK2 mutation carriers. PLoS One. 2017 Apr 13;12(4):e0175424. doi: 10.1371/journal.pone.0175424. eCollection 2017. PMID 28406934